CLINICAL TRIAL: NCT04712669
Title: A Phase 2, Dose-Ranging, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study of Rodatristat Ethyl in Patients With Pulmonary Arterial Hypertension
Brief Title: A Study of Rodatristat Ethyl in Patients With Pulmonary Arterial Hypertension (Core OLE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Altavant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RVT-1201-2002 / ELEVATE 2
Record Dates: First submitted 2021-01-12; First posted 2021-01-15 (Actual); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — rodatristat; BID protein, human

STUDY DESIGN:
Intervention Model Description: Following screening assessments, Patients will be enrolled into 1 of 3 treatment arms in a core double blind phase in 1:1:1 randomization. Subjects are allowed to participant into open label extension phase upon completion of double blind phase.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Rodatristat Ethyl 300 mg BID (Experimental): MAIN study: Rodatristat ethyl 300 mg and placebo tablet BID + standard of care medication(s) taken for 24 weeks
  Interventions: Drug: rodatristat ethyl 300 mg tablet BID
- Rodatristat Ethyl 600 mg BID (Experimental): MAIN study:Rodatristat ethyl two 300 mg tablets BID + standard of care medication(s) taken for 24 weeks
  Interventions: Drug: rodatristat ethyl 600 mg BID
- Placebo (Placebo Comparator): MAIN study: Matching two placebo tablets BID+ standard of care medication(s) taken for 24 weeks
  Interventions: Drug: Placebo
- Placebo-Rodatristat Ethyl 300 mg (Experimental): Subjects whose actual treatment group is Placebo in the double-blind phase (Main Study) and received Rodatristat ethyl two 300 mg tablets BID in the open-label phase
  Interventions: Drug: rodatristat ethyl 300 mg tablet BID
- Placebo-Rodatristat Ethyl 600 mg (Experimental): Subjects whose actual treatment group is Placebo in the double-blind phase (Main Study) and received Rodatristat ethyl two 600 mg tablets BID in the open-label phase
  Interventions: Drug: rodatristat ethyl 600 mg BID
- Rodatristat Ethyl 300 mg-Rodatristat Ethyl 300 mg (Experimental): Subjects whose actual treatment group is Rodatristat ethyl two 300 mg in the double-blind phase (Main Study) and received Rodatristat ethyl two 300 mg tablets BID in the open-label phase
  Interventions: Drug: rodatristat ethyl 300 mg tablet BID
- Rodatristat Ethyl 300 mg-Rodatristat Ethyl 600 mg (Experimental): Subjects whose actual treatment group is Rodatristat ethyl two 300 mg in the double-blind phase (Main Study) and received Rodatristat ethyl two 600 mg tablets BID in the open-label phase
  Interventions: Drug: rodatristat ethyl 600 mg BID
- Rodatristat Ethyl 600 mg-Rodatristat Ethyl 600 mg (Experimental): Subjects whose actual treatment group is Rodatristat ethyl two 600 mg in the double-blind phase (Main Study) and received Rodatristat ethyl two 600 mg tablets BID in the open-label phase
  Interventions: Drug: rodatristat ethyl 600 mg BID

INTERVENTIONS:
Drug: rodatristat ethyl 300 mg tablet BID — rodatristat ethyl 300 mg tablet + matching placebo tablet twice daily on top of standard of care
  Arms: Placebo-Rodatristat Ethyl 300 mg; Rodatristat Ethyl 300 mg BID; Rodatristat Ethyl 300 mg-Rodatristat Ethyl 300 mg
Drug: rodatristat ethyl 600 mg BID — 2 rodatristat ethyl 300 mg tablets twice daily on top of standard of care
  Arms: Placebo-Rodatristat Ethyl 600 mg; Rodatristat Ethyl 300 mg-Rodatristat Ethyl 600 mg; Rodatristat Ethyl 600 mg BID; Rodatristat Ethyl 600 mg-Rodatristat Ethyl 600 mg
Drug: Placebo — 2 matching placebo tablets on top of standard of care
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Rodatristat Ethyl in pulmonary arterial hypertension (PAH) patients.

DETAILED DESCRIPTION:
Rodatristat Ethyl is a peripherally restricted TPH inhibitor being studied as a potential treatment for PAH. This dose-ranging, randomized, double-blind, placebo-controlled, multicenter study will evaluate the effect of Rodatristat Ethyl from baseline on pulmonary vascular resistance as measured at right heart catheterization.

Patients will be enrolled into a main study with an option to enroll into an open label extension.

The study is expected to enroll patients in the USA, Canada and Europe.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female 18 years or older 2. Body Mass Index (BMI) >18kg/m2 to <=40kg/m2 3. Symptomatic PAH belonging to one of the following 2018 WHO Clinical Group 1 subtypes:

a. Idiopathic PAH b. Heritable PAH c. Drug- or toxin-induced d. PAH associated with:

1. Connective tissue disease
2. Congenital systemic to pulmonary shunt (atrial septal defect, ventricular septal defect, patent ductus arteriosus) repaired at least one year prior to Screening
3. Human immunodeficiency virus (HIV) infection - if diagnosed with HIV, must have stable disease status defined as follows:

   1. stable treatment with HIV medications for at least 8 weeks prior to Screening
   2. no active opportunistic infection during the Screening Period
   3. no hospitalizations due to HIV for at least 4 weeks prior to Screening
4. WHO FC II or III
5. Confirmed diagnosis of PAH and meet all the following hemodynamic criteria by means of a screening RHC completed prior to randomization:

   1. mPAP of >20 mmHg
   2. PVR ≥ 350 dyne•sec/cm5
   3. Pulmonary capillary wedge pressure (PCWP) or left ventricular end diastolic pressure (LVEDP) of ≤ 12 mmHg if PVR ≥ 350 and < 500 dyne•sec/cm5, or PCWP/LVEDP ≤ 15 mmHg if PVR ≥ 500 dyne•sec/cm5
6. 6MWD of 100 to 550 meters at Screening
7. Currently on a stable treatment regimen with one or more treatments approved for PAH. Stable therapy is defined as receiving the same medication(s) for ≥ 12 weeks prior to the screening RHC and at a stable dose level for each for ≥ 8 weeks prior to the screening RHC (see Protocol Section 6.6.2 for approved PAH medications). Any instances where doses of a medication have been missed prior to RHC must be discussed with the Medical Monitor prior to performing the RHC.
8. Meet all of the following criteria determined by pulmonary function tests completed no more than 24 weeks prior to Screening (performed with or without bronchodilation):

   1. Forced expiratory volume in one second (FEV1) ≥ 60% of predicted normal, and
   2. Total lung capacity (TLC) ≥ 70% of predicted normal or FVC ≥ 70% predicted if TLC is not available; For subjects with CTD associated PAH, if TLC is ≥ 60% of predicted but < 70% of predicted of if FVC ≥ 60% or predicted but < 70% of predicted, high resolution computed tomography [HRCT] obtained within 6 months of screening may be utilized to demonstrate limited interstitial lung disease
9. If participating in an exercise program for pulmonary rehabilitation, the program must have been initiated ≥ 12 weeks prior to Screening, and patient must agree to maintain the current level of rehabilitation for the first 24 weeks of receiving IP. If not participating in an exercise training program for pulmonary rehabilitation, patient must agree not to enroll in an exercise training program for pulmonary rehabilitation during the Screening Period and the first 24 weeks of receiving IP.

Exclusion Criteria:

1. Women of childbearing potential who are pregnant, planning to become pregnant, or lactating or female/male patients unwilling to use effective contraception
2. WHO pulmonary hypertension (PH) Group 1 PAH associated with portal hypertension or schistosomiasis; PH due to left heart disease (WHO PH Group 2), lung diseases and/or hypoxia (WHO PH Group 3), chronic thromboembolic PH (WHO PH Group 4), or PH with unclear multifactorial mechanisms (WHO PH Group 5)
3. PH associated with significant venous or capillary involvement (PCWP > 15 mmHg), pulmonary capillary hemangiomatosis, portal hypertension, or unrepaired congenital heart defects (CHD)
4. Three or more of the following risk factors for left ventricular disease:

   1. BMI > 30 kg/m2
   2. Diagnosis of essential hypertension that is actively treated
   3. Diabetes mellitus
   4. History of significant coronary artery disease (e.g., chronic stable angina, history of coronary intervention within the last 3 months, or a stenosis > 70% at coronary angiography)
   5. Atrial fibrillation
   6. Left atrial volume index > 41 mL/m2 [or left atrial diameter (LA) > 4 cm if LAVi unavailable]
5. Known genetic hypertrophic cardiomyopathy
6. Known cardiac sarcoidosis or amyloidosis
7. The patient has a history of, or currently has, a constrictive cardiomyopathy.
8. Known history of any left ventricular ejection fraction (LVEF) < 40% by echocardiogram within 3 years of randomization (Note: a transient decline in LVEF below 40% that occurred and recovered more than 6 months before the start of Screening and was associated with an acute intercurrent condition [e.g., atrial fibrillation] is allowed).
9. Hemodynamically significant valvular heart disease as determined by the Investigator, including:

   1. greater than mild aortic and/or mitral stenosis and/or
   2. severe mitral and/or aortic regurgitation (> Grade 3)
10. Severe arthritis, musculoskeletal problems, or morbid obesity that, in the opinion of the Investigator, is the cause of the patient's functional limitation and would affect the patient's ability to perform or complete the 6MWT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard M Lazarus, MD, FCCP, Study Director — Altavant Sciences GmbH
Locations (64):
- United States (28):
  - Arizona Pulmonary Specialists, Phoenix, Arizona
  - University of California San Diego Health Sciences, La Jolla, California
  - VA Greater LA Healthcare System/UCLA, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - Jeffrey S. Sager, MD Medical Corporation, Santa Barbara, California
  - University of Colorado, Aurora, Colorado
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Mayo Clinic Florida, Jacksonville, Florida
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Norton Pulmonary Specialists, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital (BWH), Harvard Medical School, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of New Mexico Heath Science Center, Albuquerque, New Mexico
  - NYU Langone Health, New York, New York
  - University of Rochester, Rochester, New York
  - University of North Carolina Medical Center - Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Physicians, Cincinnati, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Brown University - Rhode Island Hospital, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
- Austria (2):
  - Ordensklinikum Linz GmbH Elisabethinen, Linz, Upper Austria
  - AKH- Wien, Medizinische Univsersität Wien, Vienna
- Belgium (2):
  - Hôpital Erasme, Brussels, Brussels Capital
  - UZ Leuven - Campus Gasthuisberg - Pneumologie, Leuven, Vlaams Brabant
- Bosnia and Herzegovina (2):
  - University Clinical Centre of the Republic of Srpska, Banja Luka
  - University Clinical Hospital Mostar, Mostar
- University MHAT "Sv. Anna", Sofia, Sofia-Grad, Bulgaria
- Canada (4):
  - Peter Lougheed Centre, Calgary, Alberta
  - London Health Sciences Centre - Victoria Hospital, London, Ontario
  - University Health Network, Toronto General Hospital, Toronto, Ontario
  - Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec
- Czechia (2):
  - Fakultni nemocnice Olomouc, Olomouc
  - Vseobecna fakultni nemocnice v Praze, Prague
- France (4):
  - Centre Hospitalier Universitaire (CHU) de Caen - Hopital Cote de Nacre, Caen, Calvados
  - Groupement Hospitalier Est, Lyon, Rhône
  - Chu De Bicetre, Le Kremlin-Bicêtre, Val-de-Marne
  - CHU de Saint-Etienne - Hopital Nord, Saint-Etienne
- Universitätsklinikum Giessen und Marburg, Giessen, Germany
- Italy (3):
  - Umberto I Policlinico di Roma, Università La Sapienza, Rome, Roma
  - AOU S.Martino, IRCCS, IST-Istituto Nazionale Ricerca Sul Can, Genova
  - IRCCS Policlinico San Matteo, Università degli studi di Pavi, Pavia
- P.Stradina Clinical University Hospital, Riga, Latvia
- Spitalul Clinic Republican, Chisinau, Moldova
- Poland (4):
  - Wojewodzki Specjalistyczny Szpital im. dr Wl. Bieganskiego, Lodz, Lódzkie
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Samodzielny Publiczny Szpital Kliniczny nr 4 w Lublinie, Lublin
  - Europejskie Centrum Zdrowia Otwock Szpital im Fryderyka Chopina, Otwock
- Serbia (3):
  - Institute for Cardiovascular diseases of Vojvodina, Kamenitz, Vojvodina
  - Institute for Pulmonary Diseases of Vojvodina, Kamenitz, Vojvodina
  - Clinical Center of Serbia, Belgrade
- Spain (2):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- Ukraine (2):
  - Dnipropetrovsk Regional Clinical Diagnostic Center, Dnipro, Dnipropetrovsk Oblast
  - Nats Naukovyi Tsentr Amn Ukrainy, Kyiv
- United Kingdom (2):
  - Royal Free London NHS Foundation Trust, London
  - Royal Brompton Hospital, London

REFERENCES:
- [Derived] Sitbon O, Skride A, Feldman J, Sahay S, Shlobin OA, McLaughlin V, Ghofrani HA, Langleben D, Parsley E, D'Souza G, Marmon T, Kamau-Kelley W, Jones R, Grewal R, Wring S, Palacios M, Naik H, Denning J, Lazarus HM, Humbert M. Safety and efficacy of rodatristat ethyl for the treatment of pulmonary arterial hypertension (ELEVATE-2): a dose-ranging, randomised, multicentre, phase 2b trial. Lancet Respir Med. 2024 Nov;12(11):865-876. doi: 10.1016/S2213-2600(24)00226-1. Epub 2024 Sep 19. PMID 39307144

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 108 subjects who are dosed in Double Blind phase 76 Subjects have enrolled in Open Label extension phase.
Period: Double Blind Phase
Arm/Group | Rodatristat Ethyl 300 mg BID | Rodatristat Ethyl 600 mg BID | Placebo | Placebo-Rodatristat Ethyl 300 mg | Placebo-Rodatristat Ethyl 600 mg | Rodatristat Ethyl 300 Mg-Rodatristat Ethyl 300 mg | Rodatristat Ethyl 300 Mg-Rodatristat Ethyl 600 mg | Rodatristat Ethyl 600 Mg-Rodatristat Ethyl 600 mg
Started | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0
Completed | 28 | 26 | 32 | 0 | 0 | 0 | 0 | 0
Not Completed | 8 | 10 | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 4 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Termination by Sponsor | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Open Label Phase
Arm/Group | Rodatristat Ethyl 300 mg BID | Rodatristat Ethyl 600 mg BID | Placebo | Placebo-Rodatristat Ethyl 300 mg | Placebo-Rodatristat Ethyl 600 mg | Rodatristat Ethyl 300 Mg-Rodatristat Ethyl 300 mg | Rodatristat Ethyl 300 Mg-Rodatristat Ethyl 600 mg | Rodatristat Ethyl 600 Mg-Rodatristat Ethyl 600 mg
Started | 0 | 0 | 0 | 15 | 16 | 22 | 2 | 21
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 15 | 16 | 22 | 2 | 21
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 2
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 5 | 5 | 0 | 4
Not completed — Termination by Sponsor | 0 | 0 | 0 | 11 | 9 | 14 | 0 | 14

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Rodatristat Ethyl 300 mg BID | Rodatristat Ethyl 600 mg BID | Placebo | Placebo-Rodatristat Ethyl 300 mg | Placebo-Rodatristat Ethyl 600 mg | Rodatristat Ethyl 300 Mg-Rodatristat Ethyl 300 mg | Rodatristat Ethyl 300 Mg-Rodatristat Ethyl 600 mg | Rodatristat Ethyl 600 Mg-Rodatristat Ethyl 600 mg | Total
Number analyzed (Participants) | 36 | 36 | 36 | 15 | 16 | 22 | 2 | 21 | 184
Age, Categorical [Count of Participants; unit: Participants] — Population: Safety Population
  Participants
    Double Blind Phase: number analyzed (Participants) | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 108
    Double Blind Phase: <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Double Blind Phase: Between 18 and 65 years | 22 | 29 | 27 | 0 | 0 | 0 | 0 | 0 | 78
    Double Blind Phase: >=65 years | 14 | 7 | 9 | 0 | 0 | 0 | 0 | 0 | 30
    Open Label Phase: number analyzed (Participants) | 0 | 0 | 0 | 15 | 16 | 22 | 2 | 21 | 76
    Open Label Phase: <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Open Label Phase: Between 18 and 65 years | 0 | 0 | 0 | 10 | 13 | 10 | 2 | 16 | 51
    Open Label Phase: >=65 years | 0 | 0 | 0 | 5 | 3 | 12 | 0 | 5 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Safety Population
  Years
    Double Blind Phase: number analyzed (Participants) | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 108
    Double Blind Phase | 56.4 (14.3) | 48.4 (15.31) | 53.7 (13.76) |  |  |  |  |  | 52.83 (14.84)
    Open Label Phase: number analyzed (Participants) | 0 | 0 | 0 | 15 | 16 | 22 | 2 | 21 | 76
    Open Label Phase |  |  |  | 53.8 (13.96) | 53.4 (14.19) | 59.8 (15.84) | 53.0 (5.65) | 51.1 (13.3) | 54.68 (14.65)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Safety Population
  Participants
    Double Blind Phase: number analyzed (Participants) | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 108
    Double Blind Phase: Female | 28 | 31 | 26 | 0 | 0 | 0 | 0 | 0 | 85
    Double Blind Phase: Male | 8 | 5 | 10 | 0 | 0 | 0 | 0 | 0 | 23
    Open Label Phase: number analyzed (Participants) | 0 | 0 | 0 | 15 | 16 | 22 | 2 | 21 | 76
    Open Label Phase: Female | 0 | 0 | 0 | 13 | 12 | 17 | 1 | 19 | 62
    Open Label Phase: Male | 0 | 0 | 0 | 2 | 4 | 5 | 1 | 2 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Safety Population
  Participants
    Double Blind Phase: number analyzed (Participants) | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 108
    Double Blind Phase: Hispanic or Latino | 4 | 5 | 2 | 0 | 0 | 0 | 0 | 0 | 11
    Double Blind Phase: Not Hispanic or Latino | 32 | 29 | 33 | 0 | 0 | 0 | 0 | 0 | 94
    Double Blind Phase: Unknown or Not Reported | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 3
    Open Label Phase: number analyzed (Participants) | 0 | 0 | 0 | 15 | 16 | 22 | 2 | 21 | 76
    Open Label Phase: Hispanic or Latino | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 2 | 6
    Open Label Phase: Not Hispanic or Latino | 0 | 0 | 0 | 14 | 14 | 20 | 2 | 18 | 68
    Open Label Phase: Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Safety Population
  Participants
    Double Blind Phase: number analyzed (Participants) | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 108
    Double Blind Phase: American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Double Blind Phase: Asian | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 4
    Double Blind Phase: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Double Blind Phase: Black or African American | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 3
    Double Blind Phase: White | 29 | 29 | 25 | 0 | 0 | 0 | 0 | 0 | 83
    Double Blind Phase: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Double Blind Phase: Unknown or Not Reported | 5 | 5 | 7 | 0 | 0 | 0 | 0 | 0 | 17
    Open Label Phase: number analyzed (Participants) | 0 | 0 | 0 | 15 | 16 | 22 | 2 | 21 | 76
    Open Label Phase: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
    Open Label Phase: Asian | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 4
    Open Label Phase: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Open Label Phase: Black or African American | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
    Open Label Phase: White | 0 | 0 | 0 | 11 | 10 | 17 | 2 | 17 | 57
    Open Label Phase: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Open Label Phase: Unknown or Not Reported | 0 | 0 | 0 | 3 | 3 | 3 | 0 | 3 | 12
Region of Enrollment [Count of Participants; unit: Participants] — Study participants count by region of enrollment in Double Blind Phase Population: Safety Population
  Participants
    United States: number analyzed (Participants) | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 108
    United States | 14 | 17 | 13 | 0 | 0 | 0 | 0 | 0 | 44
    Canada: number analyzed (Participants) | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 108
    Canada | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    Austria: number analyzed (Participants) | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 108
    Austria | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    Belgium: number analyzed (Participants) | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 108
    Belgium | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Bulgaria: number analyzed (Participants) | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 108
    Bulgaria | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    Czechia: number analyzed (Participants) | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 108
    Czechia | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
    France: number analyzed (Participants) | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 108
    France | 3 | 4 | 5 | 0 | 0 | 0 | 0 | 0 | 12
    Germany: number analyzed (Participants) | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 108
    Germany | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 4
    Italy: number analyzed (Participants) | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 108
    Italy | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 6
    Latvia: number analyzed (Participants) | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 108
    Latvia | 6 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 12
    Poland: number analyzed (Participants) | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 108
    Poland | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
    Spain: number analyzed (Participants) | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 108
    Spain | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 5
    United Kingdom: number analyzed (Participants) | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 108
    United Kingdom | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
    Bosnia and Herzegovina: number analyzed (Participants) | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 108
    Bosnia and Herzegovina | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    Moldova: number analyzed (Participants) | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 108
    Moldova | 3 | 5 | 4 | 0 | 0 | 0 | 0 | 0 | 12
Region of Enrollment [Count of Participants; unit: Participants] — Study participants count by region of enrollment in Open Label Phase Population: Safety Population
  Participants
    United States: number analyzed (Participants) | 0 | 0 | 0 | 15 | 16 | 22 | 2 | 21 | 76
    United States | 0 | 0 | 0 | 4 | 8 | 9 | 2 | 11 | 34
    Canada: number analyzed (Participants) | 0 | 0 | 0 | 15 | 16 | 22 | 2 | 21 | 76
    Canada | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
    Austria: number analyzed (Participants) | 0 | 0 | 0 | 15 | 16 | 22 | 2 | 21 | 76
    Austria | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
    Belgium: number analyzed (Participants) | 0 | 0 | 0 | 15 | 16 | 22 | 2 | 21 | 76
    Belgium | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
    Czechia: number analyzed (Participants) | 0 | 0 | 0 | 15 | 16 | 22 | 2 | 21 | 76
    Czechia | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 3
    France: number analyzed (Participants) | 0 | 0 | 0 | 15 | 16 | 22 | 2 | 21 | 76
    France | 0 | 0 | 0 | 2 | 2 | 3 | 0 | 3 | 10
    Germany: number analyzed (Participants) | 0 | 0 | 0 | 15 | 16 | 22 | 2 | 21 | 76
    Germany | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 3
    Italy: number analyzed (Participants) | 0 | 0 | 0 | 15 | 16 | 22 | 2 | 21 | 76
    Italy | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 3
    Latvia: number analyzed (Participants) | 0 | 0 | 0 | 15 | 16 | 22 | 2 | 21 | 76
    Latvia | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 1 | 7
    Spain: number analyzed (Participants) | 0 | 0 | 0 | 15 | 16 | 22 | 2 | 21 | 76
    Spain | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
    Bosnia and Herzegovina: number analyzed (Participants) | 0 | 0 | 0 | 15 | 16 | 22 | 2 | 21 | 76
    Bosnia and Herzegovina | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
    Moldova: number analyzed (Participants) | 0 | 0 | 0 | 15 | 16 | 22 | 2 | 21 | 76
    Moldova | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 4 | 10
Duration since PAH diagnosis [Mean (Standard Deviation); unit: Year] — Population: Safety Population
  Year
    Double Blind Phase: number analyzed (Participants) | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 108
    Double Blind Phase | 6.18 (4.268) | 6.69 (4.913) | 8.65 (6.486) |  |  |  |  |  | 7.17 (5.4)
    Open Label Phase: number analyzed (Participants) | 0 | 0 | 0 | 15 | 16 | 22 | 2 | 21 | 76
    Open Label Phase |  |  |  | 10.54 (5.97) | 7.39 (6.98) | 5.82 (4.86) | 8.05 (3.18) | 6.14 (4.85) | 7.22 (5.8)
Duration since PAH diagnosis category [Count of Participants; unit: Participants] — Population: Safety Population
  Participants
    Double Blind Phase: number analyzed (Participants) | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 108
    Double Blind Phase: <=5 years | 18 | 17 | 13 | 0 | 0 | 0 | 0 | 0 | 48
    Double Blind Phase: >5 years | 18 | 19 | 23 | 0 | 0 | 0 | 0 | 0 | 60
    Open Label Phase: number analyzed (Participants) | 0 | 0 | 0 | 15 | 16 | 22 | 2 | 21 | 76
    Open Label Phase: <=5 years | 0 | 0 | 0 | 2 | 8 | 14 | 0 | 10 | 34
    Open Label Phase: >5 years | 0 | 0 | 0 | 13 | 8 | 8 | 2 | 11 | 42
PAH classification [Count of Participants; unit: Participants] — Population: Safety Population
  Participants
    Double Blind Phase: number analyzed (Participants) | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 108
    Double Blind Phase: IPAH | 13 | 19 | 26 | 0 | 0 | 0 | 0 | 0 | 58
    Double Blind Phase: HPAH | 5 | 5 | 4 | 0 | 0 | 0 | 0 | 0 | 14
    Double Blind Phase: Drug or toxin | 3 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 8
    Double Blind Phase: PAH associated with connective tissue disease | 11 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 15
    Double Blind Phase: PAH associated with congenital systemic pulmonary shunt | 4 | 6 | 3 | 0 | 0 | 0 | 0 | 0 | 13
    Open Label Phase: number analyzed (Participants) | 0 | 0 | 0 | 15 | 16 | 22 | 2 | 21 | 76
    Open Label Phase: IPAH | 0 | 0 | 0 | 11 | 12 | 10 | 0 | 8 | 41
    Open Label Phase: HPAH | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 3 | 9
    Open Label Phase: Drug or toxin | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 5
    Open Label Phase: PAH associated with connective tissue disease | 0 | 0 | 0 | 1 | 0 | 7 | 1 | 2 | 11
    Open Label Phase: PAH associated with congenital systemic pulmonary shunt | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 5 | 10
Number of PAH therapies category [Count of Participants; unit: Participants] — Population: Safety Population
  Participants
    Double Blind Phase: number analyzed (Participants) | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 108
    Double Blind Phase: 1 PAH therapy | 5 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 17
    Double Blind Phase: 2 PAH therapies | 12 | 12 | 11 | 0 | 0 | 0 | 0 | 0 | 35
    Double Blind Phase: 3 PAH therapies | 19 | 18 | 19 | 0 | 0 | 0 | 0 | 0 | 56
    Open Label Phase: number analyzed (Participants) | 0 | 0 | 0 | 15 | 16 | 22 | 2 | 21 | 76
    Open Label Phase: 1 PAH therapy | 0 | 0 | 0 | 3 | 3 | 3 | 1 | 4 | 14
    Open Label Phase: 2 PAH therapies | 0 | 0 | 0 | 4 | 5 | 10 | 0 | 6 | 25
    Open Label Phase: 3 PAH therapies | 0 | 0 | 0 | 8 | 8 | 9 | 1 | 11 | 37
Baseline use of selexipag [Count of Participants; unit: Participants] — Population: Safety Population
  Participants
    Double Blind Phase: number analyzed (Participants) | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 108
    Double Blind Phase: Yes | 8 | 9 | 8 | 0 | 0 | 0 | 0 | 0 | 25
    Double Blind Phase: No | 28 | 27 | 28 | 0 | 0 | 0 | 0 | 0 | 83
    Open Label Phase: number analyzed (Participants) | 0 | 0 | 0 | 15 | 16 | 22 | 2 | 21 | 76
    Open Label Phase: Yes | 0 | 0 | 0 | 2 | 3 | 2 | 0 | 5 | 12
    Open Label Phase: No | 0 | 0 | 0 | 13 | 13 | 20 | 2 | 16 | 64
Baseline use of parenteral prostacyclin [Count of Participants; unit: Participants] — Population: Safety Population
  Participants
    Double Blind Phase: number analyzed (Participants) | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 108
    Double Blind Phase: Yes | 13 | 11 | 14 | 0 | 0 | 0 | 0 | 0 | 38
    Double Blind Phase: No | 23 | 25 | 22 | 0 | 0 | 0 | 0 | 0 | 70
    Open Label Phase: number analyzed (Participants) | 0 | 0 | 0 | 15 | 16 | 22 | 2 | 21 | 76
    Open Label Phase: Yes | 0 | 0 | 0 | 8 | 6 | 9 | 1 | 7 | 31
    Open Label Phase: No | 0 | 0 | 0 | 7 | 10 | 13 | 1 | 14 | 45
Baseline use of endothelin receptor antagonist [Count of Participants; unit: Participants] — Population: Safety Population
  Participants
    Double Blind Phase: number analyzed (Participants) | 36 | 36 | 36 | 0 | 0 | 0 | 0 | 0 | 108
    Double Blind Phase: Yes | 30 | 30 | 29 | 0 | 0 | 0 | 0 | 0 | 89
    Double Blind Phase: No | 6 | 6 | 7 | 0 | 0 | 0 | 0 | 0 | 19
    Open Label Phase: number analyzed (Participants) | 0 | 0 | 0 | 15 | 16 | 22 | 2 | 21 | 76
    Open Label Phase: Yes | 0 | 0 | 0 | 11 | 13 | 17 | 2 | 16 | 59
    Open Label Phase: No | 0 | 0 | 0 | 4 | 3 | 5 | 0 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline of Pulmonary Vascular Resistance (PVR) at Week 24
Description: Pulmonary vascular resistance (PVR) was measured by right heart catheterization (RHC)
Time Frame: 24 Weeks
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Rodatristat Ethyl 300 mg BID | Rodatristat Ethyl 600 mg BID | Placebo
Number analyzed (Participants) | 36 | 36 | 36
percent | 63.083 (18.529) | 64.219 (18.013) | 5.813 (18.052)
Statistical Analysis 1: Comparison: Rodatristat Ethyl 300 mg BID vs Placebo; Test type: Superiority; p = 0.0208, ANCOVA — LSM, SE, CIs for each treatment group; LSM Diff, SE, CIs, and p-value are estimated using an ANCOVA model incl. factors for treatment group and randomization strata with associated baseline value as a covariate; H0: The mean change from baseline in PVR at Week 24 is equal between placebo and rodatristat ethyl; Mean Difference (Final Values) = 57.27, 95% CI 2-sided [8.716 to 105.824], Standard Error of Mean 24.773
Statistical Analysis 2: Comparison: Rodatristat Ethyl 600 mg BID vs Placebo; Test type: Superiority; p = 0.0174, ANCOVA — [p-value comment as in outcome 1, analysis 1]; H0: The mean change from baseline in PVR at Week 24 is equal between placebo and rodatristat ethyl; Mean Difference (Final Values) = 58.406, 95% CI 2-sided [10.272 to 106.54], Standard Error of Mean 24.558

2. Secondary Outcome: Change From Baseline in World Health Organization (WHO) Functional Class (FC)
Description: PAH functional disease severity is classified in 4 classes (I to IV) according to World Health Organization (WHO).
  I:Patients with pulmonary hypertension (PH) but without resulting limitation of physical act.Ordinary physical act does not cause undue dyspnea,fatigue,chest pain,near syncope.
  II:Patients with PH with slight limitation of physical act.Ordinary physical act causes undue dyspnea or fatigue, chest pain,or near syncope.
  III:Patients with PH with marked limitation of physical act.Less than ordinary act causes undue dyspnea or fatigue,chest pain,or near syncope.
  IV:Patients with PH with inability to carry out any physical act without symptoms,manifest signs of right-heart failure.Dyspnea and/or fatigue may even be present at rest.Discomfort is increased by physical act
  -II, -I:Patients condition improved at WK24 compared with baseline II, I:Patients condition worsened at WK24 compared with baseline No change:Patients condition not changes at WK24 compare with baseline
Time Frame: 24 Weeks
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Rodatristat Ethyl 300 mg BID | Rodatristat Ethyl 600 mg BID | Placebo
Number analyzed (Participants) | 36 | 36 | 36
Participants
  -II | 0 | 0 | 0
  -I | 2 | 3 | 3
  No Change | 30 | 30 | 30
  I | 4 | 3 | 3
  II | 0 | 0 | 0
Statistical Analysis 1: Comparison: Rodatristat Ethyl 300 mg BID vs Placebo; Test type: Superiority; p = 0.573, Regression, Logistic — P-value based on ordinal logistic regression with treatment group and randomization stratification strata as factors at alpha=0.05; H0: The distribution of change from baseline in WHO FC at Week 24 is equal between placebo and rodatristat ethyl
Statistical Analysis 2: Comparison: Rodatristat Ethyl 600 mg BID vs Placebo; Test type: Superiority; p = 0.9911, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; H0: The distribution of change from baseline in WHO FC at Week 24 is equal between placebo and rodatristat ethyl

3. Secondary Outcome: Change From Baseline in Six-minute Walk Distance (6MWD)
Description: The six-minute walk distance (6MWD) is a simple, commonly used, standardized measure of functional exercise capacity and endurance. It is a commonly used measure of efficacy in PAH clinical studies.
Time Frame: 24 Weeks
Population: ITT population
Measure: Median (Inter-Quartile Range); unit: six-minute walk distance (6MWD) (meters)
Arm/Group | Rodatristat Ethyl 300 mg BID | Rodatristat Ethyl 600 mg BID | Placebo
Number analyzed (Participants) | 36 | 36 | 36
six-minute walk distance (6MWD) (meters) | -14.5 [-31.50 to 28.00] | 0 [-27.50 to 20.00] | 2.5 [-13.50 to 23.00]
Statistical Analysis 1: Comparison: Rodatristat Ethyl 300 mg BID vs Placebo; Test type: Superiority; p = 0.0636, Wilcoxon (Mann-Whitney) — p-value (alpha=0.05) is estimated using the aligned rank stratified Wilcoxon test with the randomization stratification factors as strata; H0: The distribution of change from baseline at Week 24 in 6MWT distance (meters) is equal between placebo and rodatristat ethyl; Median Difference (Final Values) = -33.61, 95% CI 2-sided [-69.13 to 1.91], Standard Error of Mean 18.121
Statistical Analysis 2: Comparison: Rodatristat Ethyl 600 mg BID vs Placebo; Test type: Superiority; p = 0.1573, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Median Difference (Final Values) = -19.05, 95% CI 2-sided [-45.45 to 7.35], Standard Error of Mean 13.469

4. Secondary Outcome: Change From Baseline in N-terminal Prohormone of Brain Natriuretic Peptide (NT-proBNP) Levels
Description: N-terminal prohormone of brain natriuretic peptide (NT-proBNP) is a strong predictor of disease progression and mortality in PAH patients. Current PAH treatment guidelines recommend measurement of NT-proBNP levels for both risk assessment and longitudinal follow up. NT-proBNP levels are also a good marker of response to treatment.
Time Frame: 24 Weeks
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Rodatristat Ethyl 300 mg BID | Rodatristat Ethyl 600 mg BID | Placebo
Number analyzed (Participants) | 36 | 36 | 36
pg/mL | 1145.7 (325.93) | 886.1 (275.70) | 19.8 (143.86)
Statistical Analysis 1: Comparison: Rodatristat Ethyl 300 mg BID vs Placebo; Test type: Superiority; p = 0.0014, Mixed Models Analysis; H0: The mean change from baseline at Week 24 in NT-proBNP is equal between placebo and rodatristat ethyl; Mean Difference (Final Values) = 1125.9, 95% CI 2-sided [437.39 to 1814.39], Standard Error of Mean 351.28 — Estimates from a REML MMRM with baseline covariate, fixed effects, and unstructured covariance
Statistical Analysis 2: Comparison: Rodatristat Ethyl 600 mg BID vs Placebo; Test type: Superiority; p = 0.0047, Mixed Models Analysis; H0: The mean change from baseline at Week 24 in NT-proBNP is equal between placebo and rodatristat ethyl; Mean Difference (Final Values) = 866.3, 95% CI 2-sided [265.41 to 1467.16], Standard Error of Mean 306.56 — Estimates from a REML MMRM with baseline covariate, fixed effects, and unstructured covariance

ADVERSE EVENTS:
Time Frame: Up to 48 weeks
Description: An adverse event (AE) is any untoward medical occurrence in a patient, temporally associated with the use of investigational product (IP), whether or not considered related to the IP.
Arm/Group | Rodatristat Ethyl 300 mg BID | Rodatristat Ethyl 600 mg BID | Placebo | Placebo-Rodatristat Ethyl 300 mg | Placebo-Rodatristat Ethyl 600 mg | Rodatristat Ethyl 300 Mg-Rodatristat Ethyl 300 mg | Rodatristat Ethyl 300 Mg-Rodatristat Ethyl 600 mg | Rodatristat Ethyl 600 Mg-Rodatristat Ethyl 600 mg
All-Cause Mortality (participants affected / at risk) | 1/36 | 0/36 | 0/36 | 2/15 | 0/16 | 0/22 | 0/2 | 0/21
Serious Adverse Events (participants affected / at risk) | 9/36 | 6/36 | 1/36 | 2/15 | 4/16 | 6/22 | 0/2 | 3/21
Other Adverse Events (participants affected / at risk) | 32/36 | 34/36 | 27/36 | 12/15 | 15/16 | 12/22 | 2/2 | 17/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rodatristat Ethyl 300 mg BID (N=36) | Rodatristat Ethyl 600 mg BID (N=36) | Placebo (N=36) | Placebo-Rodatristat Ethyl 300 mg (N=15) | Placebo-Rodatristat Ethyl 600 mg (N=16) | Rodatristat Ethyl 300 Mg-Rodatristat Ethyl 300 mg (N=22) | Rodatristat Ethyl 300 Mg-Rodatristat Ethyl 600 mg (N=2) | Rodatristat Ethyl 600 Mg-Rodatristat Ethyl 600 mg (N=21)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related thrombosis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anticoagulation drug level below therapeutic (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transplant evaluation (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device extrusion (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device breakage (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rodatristat Ethyl 300 mg BID (N=36) | Rodatristat Ethyl 600 mg BID (N=36) | Placebo (N=36) | Placebo-Rodatristat Ethyl 300 mg (N=15) | Placebo-Rodatristat Ethyl 600 mg (N=16) | Rodatristat Ethyl 300 Mg-Rodatristat Ethyl 300 mg (N=22) | Rodatristat Ethyl 300 Mg-Rodatristat Ethyl 600 mg (N=2) | Rodatristat Ethyl 600 Mg-Rodatristat Ethyl 600 mg (N=21)
COVID-19 (Infections and infestations) | 5 (5) | 3 (3) | 8 (8) | 3 (5) | 7 (8) | 5 (5) | 1 (1) | 6 (6)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection bacterial (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Dizziness (Nervous system disorders) | 3 (3) | 3 (3) | 5 (5) | 2 (2) | 1 (1) | 2 (2) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 3 (4) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Syncope (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anosmia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hypotonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2) | 4 (6) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 9 (11) | 17 (24) | 4 (5) | 2 (3) | 6 (11) | 1 (2) | 0 (0) | 3 (4)
Nausea (Gastrointestinal disorders) | 11 (14) | 13 (17) | 3 (4) | 3 (3) | 3 (3) | 4 (4) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (5) | 8 (9) | 0 (0) | 2 (3) | 5 (7) | 2 (3) | 0 (0) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Fatigue (General disorders) | 5 (5) | 2 (3) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 3 (3) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 4 (6) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (6) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related thrombosis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lithiasis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 14 (26) | 11 (20) | 0 (0) | 4 (10) | 7 (18) | 3 (7) | 0 (0) | 3 (6)
Aspartate aminotransferase increased (Investigations) | 5 (6) | 4 (5) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4) | 3 (4) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Anticoagulation drug level below therapeutic (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Blood pH increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic enzymes increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Essential hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Congestive hepatopathy (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.

DOCUMENTS (2):
  • Study Protocol (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/69/NCT04712669/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-28): https://cdn.clinicaltrials.gov/large-docs/69/NCT04712669/SAP_001.pdf